CLINICAL TRIAL: NCT00766714
Title: The Efficacy of the Embryo Transfer Catheter in IVF and ICSI is Operator-Dependent: a Randomized Clinical Trial
Brief Title: Efficacy Study of the Embryo Transfer Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Petra De Sutter, University Hospital Ghent
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: UZGhent 002
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2008-10-06 (Estimated); Status verified 2008-10

CONDITIONS: Infertility (IVF Patients)
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Cook K-SOFT-5100 catheter
  Interventions: Device: Cook K-SOFT-5100 catheter
- 2 (Active Comparator): Frydman classical catheter
  Interventions: Device: Frydman classical catheter

INTERVENTIONS:
Device: Cook K-SOFT-5100 catheter — A Cook K-SOFT-5100 catheter was used for embryo transfer in human IVF/ICSI
  Arms: 1
Device: Frydman classical catheter — A Frydman classical catheter was used for embryo transfer in human IVF/ICSI
  Arms: 2

SUMMARY:
A prospective randomized trial comparing Cook K-SOFT-5100 and Frydman classical catheter 4.5 for embryo transfer in human IVF/ICSI was performed. Three experienced operators participated in the trial, using a fixed distance transfer protocol. Primary endpoint was clinical pregnancy rate, secondary endpoints were rates of difficult transfer and of catheter failure. Patients were randomized by a computer program immediately prior to embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing embryo transfer in our IVF program between 2000 and 2005

Exclusion Criteria:

* patients not giving consent were excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1446 (Actual)
Dates: Start 2000-01; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rates | End of study

SECONDARY OUTCOMES:
Rates of difficult transfer | End of study
Catheter failure rate | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Petra De Sutter, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- [Derived] Yao Z, Vansteelandt S, Van der Elst J, Coetsier T, Dhont M, De Sutter P. The efficacy of the embryo transfer catheter in IVF and ICSI is operator-dependent: a randomized clinical trial. Hum Reprod. 2009 Apr;24(4):880-7. doi: 10.1093/humrep/den453. Epub 2008 Dec 18. PMID 19095665
- See also: Website of the University Hospital Ghent — http://www.uzgent.be